CLINICAL TRIAL: NCT03016455
Title: B Cell Lymphocyte in Humoral Rejection and Alloimmunisation
Acronym: BHL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: BHL (RB 12.047)
Record Dates: First submitted 2016-08-30; First posted 2017-01-10 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-04

CONDITIONS: Renal Transplant
Keywords: Kidney Transplant; Immunology
MeSH Terms: interventions — 2-methyl-3-hydroxybutyryl-coenzyme A dehydrogenase

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood

GROUPS / COHORTS (3):
- DSA positive patients without cAMR: Presence of DSA w/o cAMR
  Interventions: Other: Presence of DSA w/o cAMR
- DSA positive patients with cAMR: Presence of DSA w/ cAMR
  Interventions: Other: Presence of DSA w/ cAMR
- Stable patients: No DSA No cAMR
  Interventions: Other: No DSA No cAMR

INTERVENTIONS:
Other: Presence of DSA w/ cAMR
  Groups: DSA positive patients with cAMR
Other: Presence of DSA w/o cAMR
  Groups: DSA positive patients without cAMR
Other: No DSA No cAMR
  Groups: Stable patients

SUMMARY:
This study aims to better characterise B cell phenotype and functional abnormalities in kidney transplant patients producing donor specific antibody (DSA) and in those with chronic antibody mediated rejection (cAMR) and to search for a predictive tool (biomarker). The functional analysis will help to better understand B cell-dependant mechanisms implied in T cell proliferation and better target future treatments.

DETAILED DESCRIPTION:
The principal objective is to better understand the B cell dependant mechanisms of the chronic antibody mediated rejection (cAMR). A particular focus will be done on the mechanisms that could explain the natural history of chronic humoral mediated rejection and of pathways from DSA negative status toward DSA positive status and from DSA positive status to histological lesions. The following will be undergone for three categories of patients (stable patients, DSA positive patients without cAMR and DSA positive patients with cAMR) :

* A phenotypic analysis of B cells of patients suffering from chronic humoral rejection or who are simply DSA positive.
* A functional analysis in autologous cultures in order to confirm our preliminary results.
* A functional analysis in a heterologous proliferation test aiming at a better understanding of the absence of B cell regulation of T cell proliferation in patients suffering from cAMR.
* A cytokine analysis (IL10, alpha-tumor necrosis factor, gamma-interferon dosing), for a better understanding of the mechanisms that are involved in the regulation of the T cell response that is induced by the B cells.

ELIGIBILITY:
Inclusion criteria :

* Non stable patients :

  * Patient older than 18 years old.
  * Patient which is the recipient of a renal transplant
  * Patient who develops anti donor antibodies after the transplantation and / or suffering from a histologically-proven antibody mediated rejection.
  * Patient who has signed an informed consent form
* Stable patients :

  * Patient older than 18 years old.
  * Patient that is the recipient of a renal transplant for more than one year
  * Patient who has accepted to participate in the Brest Kidney graft recipient collection
  * Patient that is not suffering from any rejection, that has a good renal function and a low proteinuria
  * Patient that has not developed any DSA.

Exclusion criteria :

- Patients that has not signed the consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 kidney graft recipients with DSA or cAMR (renal dysfunction, positive DSA, allograft nephropathy), and 25 stable patients of 13 French transplantation centres.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2013-06; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the ratio (percentage and absolute values) of mature LB subpopulations (LBm1 to LBm5) and of memory LB by specific labellings | At the inclusion day
Evaluation of the proliferation of freshly isolated cells T in presence of autologous B cells | At the inclusion day
Evaluation of the proliferation of T cells in a heterologous test | At the inclusion day
  aiming at a better understanding of the absence of B cell regulation of T cell proliferation in patients suffering from cAMR
cytokine analysis(IL10, alpha-Tumor Necrosis FActor, gamma-Interferon dosing) | At the inclusion day
  for a better understanding of the mechanisms that are involved in the regulation of the T cell response that is induced by the B cells.

SECONDARY OUTCOMES:
Correlation between phenotypic and functional evaluations, and clinical outcome | One year post inclusion
comparison of the B cell subpopulations before and after rituximab treatment | One year post inclusion
  In a subgroup of patients, the ones that will happen to be treated by rituximab for a rejection episode.

CONTACTS AND LOCATIONS:
Overall Officials: Yannick LE MEUR, MD PhD, Study Director — University Hospital, Brest
Locations (13):
- France (13):
  - CHU Amiens, Amiens
  - Chu Angers, Angers
  - CHU Brest, Brest
  - CHU CAEN, Caen
  - Chu Clermont Ferrand, Clermont-Ferrand
  - CHU Limoges, Limoges
  - APHP Hôpital Necker, Paris
  - CHU Poitiers, Poitiers
  - CHU Reims, Reims
  - CHU Rennes, Rennes
  - CHU Rouen, Rouen
  - Hôpitaux Universitaires de Strasbourg, Strasbourg
  - CHU Tours, Tours